CLINICAL TRIAL: NCT05884671
Title: Dopaminergic Mechanisms of Gating Working Memory, Learning and Motivation: a Pharmaco-fMRI Study
Brief Title: Dopamine and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donders Centre for Cognitive Neuroimaging (Other)
Collaborators: Prof. Dr. Robbert-Jan Verkes, Radboud University Medical Centre Department of Psychiatry (Unknown); Funding: NWO + KNAW (Unknown)
Responsible Party: Principal Investigator, Roshan Cools, Prof. Dr., Donders Centre for Cognitive Neuroimaging
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 3017048.09
Record Dates: First submitted 2023-03-21; First posted 2023-06-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Sulpiride's Effect on Striatal BOLD Signal During Working Memory Gating; Interaction of Sulpiride, Average Reward Rate and Evidence Accumulation; Interaction of Sulpiride, Average Reward Rate and Cognitive Effort
MeSH Terms: interventions — Sulpiride

STUDY DESIGN:
Intervention Model Description: This is a within-subjects (i.e., crossover), double-blind, randomized placebo-controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulpiride (Active Comparator): All study participants receive both placebo and the active medication (sulpiride 400mg), in a within-subjects , double-blind, randomized design.
  Interventions: Drug: Sulpiride 400 MG
- Placebo (Placebo Comparator): All study participants receive both placebo and the active medication (sulpiride 400mg), in a within-subjects , double-blind, randomized design.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulpiride 400 MG — All participants will receive one single dose of 400mg sulpiride. None of the participants will receive repeated doses. In order for the fMRI data acquisition to coincide with the time-window of maximal drug effects represented by a combination of plasma kinetics and physiological effects we will administer the drug 90 minutes prior to fMRI data acquisition.
  Other Names: Dogmatil
  Arms: Sulpiride
Drug: Placebo — All participants will receive placebo during one of the sessions.
  Arms: Placebo

SUMMARY:
Rationale: To unravel the role of dopamine in gating of working memory, motivation and learning.

Objective: The primary objective of this study is to isolate effects of blocking D2 receptor stimulation on gating of working memory, reinforcement learning and reward-based motivation, and their associated physiological changes (measured with fMRI and eye tracking). The secondary objective is to assess the degree to which the effects of D2 receptor action vary as a function of proxy measures of baseline dopamine levels.

Study design: A double-blind placebo controlled within-subject design will be employed, in which young healthy participants are tested twice, once on placebo, and once on a low oral dose (400mg) of the D2 receptor antagonist sulpiride. This design and drug dose is commonly used in our lab without side effects (previously approved CMO protocols 2011/204, 2008/078 & 2016/2646).

Study population: Healthy human participants, 18 - 45 yr old. We will recruit 46 participants.

Intervention: Participants will receive both 400 mg sulpiride and placebo, in separate sessions in a counterbalanced order.

Main study parameters/endpoints: BOLD signal measured with fMRI, and behavioural performance on cognitive tasks.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will attend 3 study sessions: A screening session and 2 pharmaco-fMRI sessions (sulpiride and placebo). Participants will complete a baseline battery of tasks and questionnaires, a structural MRI scan, as well as a battery of tasks both in and outside the scanner. On the day preceding each pharmaco-fMRI session, participants will have to adhere to some simple restrictions with respect to medication, alcohol and drug intake. On the day of testing participants will have to refrain from smoking and stimulant-containing drinks. Sulpiride can be administered safely without any relevant risk of serious adverse events and has been approved for clinical use in the Netherlands.

DETAILED DESCRIPTION:
A more detailed description can be found in the approved research protocol as well as the pre-registrations. The links to the pre-registrations will be made available upon publication.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 45 years of age
* Predominant right-handedness

Exclusion Criteria:

* Presence of prolactin-dependent tumors (e.g., pituitary prolactinoma or breast cancer)
* (History of) autonomic failure (e.g., vasovagal reflex syncope).
* (History of) clinically significant hepatic, cardiac, obstructive respiratory, renal, cerebrovascular, cardiovascular, metabolic, ocular or pulmonary disease/disorders
* (History of) epilepsy in adulthood (i.e. no insult after 18 years of age, no current medication for epilepsy and no insult in the last five years)
* Diagnosis (or history of) endocrine treatment
* Diagnosis (or history of) neuroendocrine treatment (e.g., phechromocytoma, hyperthyroidism, Cushing's syndrome)
* (History of) melanoma
* Hypersensitivity to sulpiride
* One first degree or two or more second degree family members with a history of sudden death or ventricular arrhythmia
* Abnormal QT interval (assessed via ECG)
* Uncontrolled hypertension, defined as diastolic blood pressure at rest > 95 mmHg or systolic blood pressure at rest > 180 mmHg
* Hypotension, defined as diastolic blood pressure < 50 mm Hg or systolic < 95 mm Hg
* or resting pulse rate < 45 beats/min
* Diabetes
* History of prescribed medication within the last month prior to the start of the study.
* History of 'over the counter' medication within the last two months (with exception of occasional use of paracetamol, acetylsalicylic acid, and ibuprofen).
* Possible pregnancy or breastfeeding
* No appropriate contraception
* Undiagnosed skin lesions
* Lactose intolerance
* Glaucoma or increased risk for glaucoma
* Possible pregnancy or breastfeeding
* Metal objects in or around the body (braces, pacemaker, metal fragments, hearing devices)
* Claustrophobia
* Diagnosis (or history of) psychiatric treatment (e.g., severe depression, anorexia nervosa, severe mood disorders, mania, schizophrenia or borderline personality disorder)
* Diagnosis (or history of) neurological treatment
* (History of) drug dependence (opiate, LSD, (meth)amphetamine, cocaine, solvents, or barbiturate) or alcohol dependence
* Suicidality
* Use of MAO inhibitor, anaesthetic, antidepressant or antipsychotic drugs within the week prior to the start of the study.
* Average use of psychotropic medication or recreational drugs weekly or more.
* Cannabis use within 2 weeks prior to the start of the study, and periods of more than 3 months using weekly or more in the last 6 months
* Use of psychotropic medication, or of recreational drugs over a period of 72 hours
* prior to the test sessions, and use of alcohol within the last 24 hours before each measurement.
* Average use of more than 3 alcohol beverages daily.
* Average use of psychotropic medication or recreational drugs weekly or more.
* Habitual smoking, i.e., more than a pack of cigarettes per week and/or a self-reported inability or unease to cease smoking for 24 hours to testing.
* Regular use of corticosteroids.
* Abnormal hearing or (uncorrected) vision.
* First degree family member with schizophrenia or bipolar disorder
* Irregular sleep/wake rhythm (e.g., regular nightshifts or cross timezone travel).
* Left handedness (because lateralisations of brain activation may differ from right-handed people).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Working memory gating task: Reaction time | Measured at intervention day 1, 115 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Reaction time [ms] during selective vs. non-selective input- and output-gating to assess the ability (speed) to selectively input- and output-gate working memory representations at intervention (sulpiride) versus placebo.
Working memory gating task: Reaction time | Measured at intervention day 2, 115 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Reaction time [ms] during selective vs. non-selective input- and output-gating to assess the ability (speed) to selectively input- and output-gate working memory representations at intervention (sulpiride) versus placebo.
Working memory gating task: Accuracy | Measured at intervention day 1, 115 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Accuracy [%] during selective vs. non-selective input- and output-gating to assess the ability (correctness) to selectively input- and output-gate working memory representations at intervention (sulpiride) versus placebo.
Working memory gating task: Accuracy | Measured at intervention day 2, 115 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Accuracy [%] during selective vs. non-selective input- and output-gating to assess the ability (correctness) to selectively input- and output-gate working memory representations at intervention (sulpiride) versus placebo.
Working memory gating task: BOLD-response | Measured at intervention day 1, 115 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  BOLD-response to selective vs. global cues, examined for both pre- and retro-cue conditions (i.e., input- and output-gating respectively) to assess the neural response to selective working memory gating at intervention (sulpiride) versus placebo.
Working memory gating task: BOLD-response | Measured at intervention day 2, 115 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  BOLD-response to selective vs. global cues, examined for both pre- and retro-cue conditions (i.e., input- and output-gating respectively) to assess the neural response to selective working memory gating at intervention (sulpiride) versus placebo.
Simon task: Accuracy | Measured at intervention day 1, 250 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Accuracy [%] during high and low average reward rate congruent and incongruent trials to assess cognitive effort investment after intervention versus placebo.
Simon task: Accuracy | Measured at intervention day 2, 250 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Accuracy [%] during high and low average reward rate congruent and incongruent trials to assess cognitive effort investment after intervention versus placebo.
Simon task: Reaction time | Measured at intervention day 1, 250 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Reaction time [ms] during high and low average reward rate congruent and incongruent trials to assess cognitive effort investment after intervention versus placebo
Simon task: Reaction time | Measured at intervention day 2, 250 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Reaction time [ms] during high and low average reward rate congruent and incongruent trials to assess cognitive effort investment after intervention versus placebo
Perceptual decision-making task: Accuracy | Measured at intervention day 1, 215 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Accuracy [%] as a function of average reward rate to assess cognitive effort investment after intervention versus placebo.
Perceptual decision-making task: Accuracy | Measured at intervention day 2, 215 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Accuracy [%] as a function of average reward rate to assess cognitive effort investment after intervention versus placebo.
Perceptual decision-making task: Reaction time | Measured at intervention day 1, 215 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Reaction time [ms] as a function of average reward rate to assess cognitive effort investment after intervention versus placebo.
Perceptual decision-making task: Reaction time | Measured at intervention day 2, 215 min after the pharmacological intervention took place. Measurements are compared regarding intervention type (drug versus placebo).
  Reaction time [ms] as a function of average reward rate to assess cognitive effort investment after intervention versus placebo.

SECONDARY OUTCOMES:
Eye-blink rate | Measured at baseline during intake session
  Number of spontaneous eye blinks per minute, as a clinically relevant biomarker of striatal dopamine function
Operation Span test | Measured at baseline during intake session
  Number of letters remembered while performing math problems, as a parameter for working memory capacity
Digit Span test | Measured at baseline during intake session
  Accuracy score [nr of correct responses] on forward span and backward span, as a parameter for working memory capacity
Digit Span test | Measured during intervention day 1 (sessions at least 14 days apart), 290 min after the pharmacological intervention took place
  Accuracy score [nr of correct responses] on forward span and backward span, as a parameter for working memory capacity
Digit Span test | Measured during intervention day 2 (sessions at least 14 days apart), 290 min after the pharmacological intervention took place
  Accuracy score [nr of correct responses] on forward span and backward span, as a parameter for working memory capacity
Beck Depression Inventory | Baseline measure via online questionnaire in between first and second intervention session (these take place at least 14 days apart)
  Average score as indicator of depressive symptoms
Barratt Impulsiveness Scale | Baseline measure via online questionnaire in between first and second intervention session (these take place at least 14 days apart)
  Average score as indicator of impulsivity (personality trait)
Behavioural Inhibition Scale/Behavioural Activation Scale | Baseline measure via online questionnaire in between first and second intervention session (these take place at least 14 days apart)
  Average score as indicator of behavioural activation and inhibition
State and Trait Anxiety Inventory | Baseline measure via online questionnaire in between first and second intervention session (these take place at least 14 days apart)
  Average score as indicator of state and trait anxiety
Utrechtse Burnout Schaal/Maslach Burnout Inventory | Baseline measure via online questionnaire in between first and second intervention session (these take place at least 14 days apart)
  Average score as indicator of burn out
Covid-19 Stress Scales | Baseline measure via online questionnaire in between first and second intervention session (these take place at least 14 days apart)
  Average score as indicator of COVID-related stress and anxiety

OTHER OUTCOMES:
Diastolic blood pressure | Measured at baseline on intervention day 1 (before pharmacological intervention took place)
  Unit of measurement: mmHG
Diastolic blood pressure | Measured at baseline on intervention day 2 (before pharmacological intervention took place)
  Unit of measurement: mmHG
Diastolic blood pressure | Measured 90 min post drug/placebo intake on intervention day 1
  Unit of measurement: mmHG
Diastolic blood pressure | Measured 90 min post drug/placebo intake on intervention day 2
  Unit of measurement: mmHG
Diastolic blood pressure | Measured 300 min post drug/placebo intake on intervention day 1
  Unit of measurement: mmHG
Diastolic blood pressure | Measured 300 min post drug/placebo intake on intervention day 2
  Unit of measurement: mmHG
Systolic blood pressure | Measured at baseline on intervention day 1 (before pharmacological intervention took place)
  Unit of measurement: mmHG
Systolic blood pressure | Measured at baseline on intervention day 2 (before pharmacological intervention took place)
  Unit of measurement: mmHG
Systolic blood pressure | Measured 90 min post drug/placebo intake on intervention day 1
  Unit of measurement: mmHG
Systolic blood pressure | Measured 90 min post drug/placebo intake on intervention day 2
  Unit of measurement: mmHG
Systolic blood pressure | Measured 300 min post drug/placebo intake on intervention day 1
  Unit of measurement: mmHG
Systolic blood pressure | Measured 300 min post drug/placebo intake on intervention day 2
  Unit of measurement: mmHG
Heart rate | Measured at baseline on intervention day 1 (before pharmacological intervention took place)
  Unit of measurement: beats per minute (bpm)
Heart rate | Measured at baseline on intervention day 2 (before pharmacological intervention took place)
  Unit of measurement: beats per minute (bpm)
Heart rate | Measured 90 min post drug/placebo intake on intervention day 1
  Unit of measurement: beats per minute (bpm)
Heart rate | Measured 90 min post drug/placebo intake on intervention day 2
  Unit of measurement: beats per minute (bpm)
Heart rate | Measured 300 min post drug/placebo intake on intervention day 1
  Unit of measurement: beats per minute (bpm)
Heart rate | Measured 300 min post drug/placebo intake on intervention day 2
  Unit of measurement: beats per minute (bpm)
Body temperature | Measured at baseline on intervention day 1 (before pharmacological intervention took place)
  Measured in degree Celsius by an in-ear thermometer
Body temperature | Measured at baseline on intervention day 2 (before pharmacological intervention took place)
  Measured in degree Celsius by an in-ear thermometer
Body temperature | Measured 90 min post drug/placebo intake on intervention day 1
  Measured in degree Celsius by an in-ear thermometer
Body temperature | Measured 90 min post drug/placebo intake on intervention day 2
  Measured in degree Celsius by an in-ear thermometer
Body temperature | Measured 300 min post drug/placebo intake on intervention day 1
  Measured in degree Celsius by an in-ear thermometer
Body temperature | Measured 300 min post drug/placebo intake on intervention day 2
  Measured in degree Celsius by an in-ear thermometer
Respiration movements | Measured during the MRI scan (115 min post drug/placebo) on intervention day 1. The pharmacological intervention sessions take place at least 14 days apart)
  Voltage change over time measured by a respiration belt around participants' abdomen during MRI scanning
Respiration movements | Measured during the MRI scan (115 min post drug/placebo) on intervention day 2. The pharmacological intervention sessions take place at least 14 days apart)
  Voltage change over time measured by a respiration belt around participants' abdomen during MRI scanning
Visual Analogue Scale (VAS) | Measured at baseline on intervention day 1 (before pharmacological intervention took place)
  Measured with 16 mood rating items measured on a continuous scale from 1 to 10 by self-report
Visual Analogue Scale (VAS) | Measured at baseline on intervention day 2 (before pharmacological intervention took place)
  Measured with 16 mood rating items measured on a continuous scale from 1 to 10 by self-report
Visual Analogue Scale (VAS) | Measured 90 min post drug/placebo intake on intervention day 1
  Measured with 16 mood rating items measured on a continuous scale from 1 to 10 by self-report
Visual Analogue Scale (VAS) | Measured 90 min post drug/placebo intake on intervention day 2
  Measured with 16 mood rating items measured on a continuous scale from 1 to 10 by self-report
Visual Analogue Scale (VAS) | Measured 300 min post drug/placebo intake on intervention day 1
  Measured with 16 mood rating items measured on a continuous scale from 1 to 10 by self-report
Visual Analogue Scale (VAS) | Measured 300 min post drug/placebo intake on intervention day 2
  Measured with 16 mood rating items measured on a continuous scale from 1 to 10 by self-report
Positive and Negative Affect Scale (PANAS) | Measured at baseline on intervention day 1 (before pharmacological intervention took place)
  Measured with 20 statements regarding feelings and emotions measured on a 5-point Likert scale by self-report
Positive and Negative Affect Scale (PANAS) | Measured at baseline on intervention day 2 (before pharmacological intervention took place)
  Measured with 20 statements regarding feelings and emotions measured on a 5-point Likert scale by self-report
Positive and Negative Affect Scale (PANAS) | Measured 90 min post drug/placebo intake on intervention day 1
  Measured with 20 statements regarding feelings and emotions measured on a 5-point Likert scale by self-report
Positive and Negative Affect Scale (PANAS) | Measured 90 min post drug/placebo intake on intervention day 2
  Measured with 20 statements regarding feelings and emotions measured on a 5-point Likert scale by self-report
Positive and Negative Affect Scale (PANAS) | Measured 300 min post drug/placebo intake on intervention day 1
  Measured with 20 statements regarding feelings and emotions measured on a 5-point Likert scale by self-report
Positive and Negative Affect Scale (PANAS) | Measured 300 min post drug/placebo intake on intervention day 2
  Measured with 20 statements regarding feelings and emotions measured on a 5-point Likert scale by self-report
Menstrual cycle stage (for female participants) | Measured within the first 10 min of the intervention day 1 (i.e., 10 min pre drug/placebo)
  Day of onset of last menstrual bleeding measured by self-report
Menstrual cycle stage (for female participants) | Measured within the first 10 min of the intervention day 2 (i.e., 10 min pre drug/placebo)
  Day of onset of last menstrual bleeding measured by self-report

CONTACTS AND LOCATIONS:
Locations (1):
- Donders Centre for Cognition, Radboud University, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Following publication, raw and processed data will be archived for scientific integrity. The data use agreement gives access to the data, provided that certain conditions set by the local institutional guidelines as well as (inter)national (EU) law are met.
  Data sharing will be done using the Donders Institute research data repository (http://data.donders.ru.nl) in accordance to institutional and EU guidelines.
Supporting Information: Analytic Code
Time Frame: After publication
Access Criteria: As described on the website of the Donders Repository, shared data can be accessed via a persistent identifier. This identifier can be obtained directly from the authors or via a link in the publication. Also see: https://data.donders.ru.nl/doc/help/user-manual/access-shared-data/request-access.html?4
URL: https://data.donders.ru.nl/